CLINICAL TRIAL: NCT01887314
Title: Multicenter, Randomized, Double-blind, Placebo Controlled, Study to Evaluate the Activity of a Ginger (Zingiber Officinale) Food Supplement in the Management of Nausea in Patients Receiving Highly Emetogenic Treatments and Standard Anti-emetogenic Therapy.
Brief Title: Efficacy Study of Ginger (Zingiber Officinale) Extract "Ginpax" to Manage Nausea in Cancer Patients Receiving High Emetogenic Treatments and Standard Anti-emetogenic Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HF01-12-69; HF01-12-69 (Other: Helsinn Healthcare SA)
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Cancer; Nausea; Vomiting
Keywords: Cancer; Cisplatin; Nausea; Ginger; Zingiber officinale; 5HT3; Dexamethasone; Neurokinin-1 (NK-1); Interleukin-6 (IL-6); Tumor necrosis factor-alpha (TNF-alpha); Insulin like growth factor-1 (IGF-1); Placebo; FLIE; BFI
MeSH Terms: conditions — Neoplasms; Nausea; Vomiting

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standardized Ginger extract soft gel capsules (Experimental): Patients receive 2 soft gel capsules of Ginger extract, twice a day
  Interventions: Dietary Supplement: Standardized Ginger extract
- Placebo soft gel capsules (Placebo Comparator): Patients receive 2 soft gel capsules of Placebo, twice a day
  Interventions: Dietary Supplement: Standardized Ginger extract

INTERVENTIONS:
Dietary Supplement: Standardized Ginger extract
  Other Names: Ginpax

SUMMARY:
The purpose of the study is verify the capability of a standardized Ginger (Zingiber officinale) extract to manage nausea in cancer patients receiving highly emetogenic treatments and standard anti-emetogenic therapy.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo controlled, multicenter study with two parallel groups of patients.

The study will be conducted in 5 Italian clinical sites and will involve 250 patients receiving at least 2 cycles of highly emetogenic treatments.

Patients will be randomly assigned to Ginger treatment or to its Placebo.

All patients will receive, at each chemotherapy cycle, the standard 5-HT3 receptor antagonist antiemetics plus dexamethasone and NK1 receptor antagonist. This will guarantee to all patients an antiemetic prophylaxis for acute and delayed nausea. No additional treatment is usually foreseen for nausea and this justifies the use of placebo in the control group.

Patients will start the study treatment on the day after chemotherapy cycle and will continue until the day of the following cycle; they will suspend the study treatment on the chemotherapy day and will start again on the next day. The choice not to treat the patients with the study product on the chemotherapy day is intended to avoid any possible interference with antiemetic therapy of the first day and chemotherapy, and to analyze the impact of Ginger in delayed phase without confounding factors in acute phase.

Main efficacy assessment of this study is:

- To evaluate the protection from delayed nausea (incidence of no delayed nausea and non-significant delayed nausea);

Other efficacy assessments regarding nausea that will be evaluated are:

* To evaluate the severity of delayed nausea;
* To evaluate the overall duration of nausea;
* To evaluate inter cycle nausea;
* To evaluate nausea anticipatory symptoms before the 2nd cycle.

Secondary efficacy assessments of this study are:

* To evaluate protection from delayed vomiting (number of emetic episodes in delayed phase);
* To evaluate the impact of nausea/vomiting on daily life activities (FLIE30 questionnaire);
* To evaluate the use of antiemetic rescue medication;
* To evaluate the compliance to the treatment;
* To assess overall fatigue (BFI31 questionnaire).

Safety assessments of this study are:

- Number and typology of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Male and Females aged > 18 years.
* Naïve to chemotherapy.
* Patients planned to receive at least 2 cycles of highly emetogenic treatments with cisplatin in single dose > 50 mg/m2 every 21 or 28 days.
* Willing and able to understand and sign informed consent and complete the patient diary.

Exclusion Criteria:

* Presence of brain symptomatic metastases (in case of small, asymptomatic metastases and in absence of steroids treatment, the patient is eligible).
* Scheduled to receive or having received in the past 4 weeks radiation treatment to brain, abdomen or pelvis.
* Emesis or significant nausea within 24 hours before first chemotherapy cycle.
* Known hypersensitivity reaction to Ginger or any components of the product.
* Patients with coagulopathies causing potential increase risk of bleeding.
* Patients on therapy with oral anticoagulants.
* Planned surgery procedures in the period of the study or within 2 weeks after the study conclusion.
* History of seizures.
* Active use of cannabinoids.
* Known current or past drug or alcohol abuse.
* Use of other investigational drugs within 30 days before study entry or during the study.
* Clinically significant findings on physical exam or presence of known clinically significant disease that would interfere with study evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2013-06; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of Ginger in protecting patients from delayed nausea (incidence of no delayed nausea and non-significant delayed nausea) | Two High Emetogenic chemotherapy cylces (41 or 55 days)
  The level of nausea will be assessed through a Visual Analogue Scale (VAS 0-100 mm) included in the patients' daily diary. The patients will be asked to report the maximum level of nausea experienced during each day.
  During each chemotherapy cycle, the nausea occurring between day 2 and day 5 will be defined as "delayed nausea", the nausea occurring between day 6 and day 19/26 will be considered as "inter-cycle nausea". The day before the next chemotherapy cycle (day 20/27), "anticipatory nausea" symptoms will be collected.

SECONDARY OUTCOMES:
Protection from delayed vomiting (number of emetic episodes in delayed phase) | Two High Emetogenic chemotherapy cylces (41 or 55 days)
Use of antiemetic rescue medication. | Two High Emetogenic chemotherapy cylces (41 or 55 days)
Overall fatigue assessment (BFI questionnaire) | Two High Emetogenic chemotherapy cylces (41 or 55 days)

OTHER OUTCOMES:
Biochemical markers | Two High Emetogenic chemotherapy cylces (41 or 55 days)
  On a restricted number of patients enrolled at the coordinating center, additional blood samples will be collected for IL-6, TNF-alpha, IGF-1 evaluation.
  The purpose of this additional research is to evaluate if the consumption of ginger can affect serum concentration of such factors.
To evaluate the safety profile of the product containing Ginger extract. | Two High Emetogenic chemotherapy cylces (41 or 55 days)
  Number and typology of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bossi, M.D., Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (6):
- Italy (6):
  - Istituto Nazionale dei Tumori, Milan
  - IEO -Istituto Europeo di Oncologia-, Milan
  - Ospedale S. Gerardo, Monza
  - Policlinico Umberto I, Rome
  - Istituti Fisioterapici Ospitalieri - Istituto Nazionale Tumori "Regina Elena", Rome
  - Ospedale S. Maria, Terni

IPD SHARING:
Plan to Share IPD: No